CLINICAL TRIAL: NCT07338994
Title: TENS With Proprioceptive-Visual Training on Gait Parameters in Children With Spastic Diplegic Cerebral Palsy: A Randomized Controlled Trial
Brief Title: TENS With Proprioceptive-Visual Training on Gait Parameters in CP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mostafa S Ali, faculty of physical therapy, cairo university, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/006102
Record Dates: First submitted 2025-12-19; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Cerebral Palsy (CP)
Keywords: Spastic diplegia; visual training; proprioceptive stimulation; gait; Tekscan Walkway; TENS
MeSH Terms: conditions — Cerebral Palsy | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Intervention Model Description: Electrical stimulation will be delivered by means of self-adherent surface electrodes (Encore plus), using a programmable electrical stimulator, providing monophasic rectangular pulse trains. Electrodes were attached over the belly of the rectus femoris and tibialis anterior muscles. The quadriceps and the dorsiflexors were selected due to their dominance in establishing a normal and efficient gait. TENS was applied for 20 minutes during gait training. The parameters selected for the electrical stimulation will be as follows: frequency 20Hz, pulse-width 0.25 msec, and intensity will be individually adjusted for each subject
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Placebo Comparator): receive proprioceptive-visual training
  Interventions: Device: 1. Tekscan Walkway system
- study group (Experimental): TENS with proprioceptive - visual training
  Interventions: Device: TENS; Device: 1. Tekscan Walkway system

INTERVENTIONS:
Device: TENS — Electrical stimulation will be delivered by means of self-adherent surface electrodes (Encore plus), using a programmable electrical stimulator, providing monophasic rectangular pulse trains. Electrodes were attached over the belly of the rectus femoris and tibialis anterior muscles. The quadriceps and the dorsiflexors were selected due to their dominance in establishing a normal and efficient gait. TENS was applied for 20 minutes during gait training. The parameters selected for the electrical stimulation will be as follows: frequency 20Hz, pulse-width 0.25 msec, and intensity will be individually adjusted for each subject
  Arms: study group
Device: 1. Tekscan Walkway system — It includes sensors (4 sensels/cm2) with a resolution of up to 185 Hz, a digital mat (195.5 cm long by 44.2 cm wide) placed in a wooden pathway, and a pressure sensor (1 to 862 kPa). The plasma screen faces the walkway and is 1.5 meters high and 7 meters away. It displays pictures that are mirrored from seven pressure points (forming the contour of the foot). if the foot's heel, midfoot, forefoot, fifth metatarsal, third-fourth, second, and first metatarsals are the seven areas of pressure. Data such as maximum peak pressure (kPa), stance time (s), cadence, gait time (s), distance (cm), velocity (cm/s), and transmission hardware (cable and sensor-interface or so-called handle) will be extrapolated using a computer running The Tekscan Software (version 7).

SUMMARY:
This study aimed to evaluate the effect of TENS with proprioceptive - visual training on gait parameters in children with spastic diplegic cerebral palsy.

DETAILED DESCRIPTION:
Two groups of thirty diplegic CP children, ages 4 to 6, were randomly assigned to receive proprioceptive-visual training as the control group and TENS with proprioceptive - visual training as the research group. For eight weeks, both groups received therapy three times a week. Prior to and during the intervention period, each participant had an evaluation by gait analysis.

ELIGIBILITY:
Inclusion Criteria:

* Diplegic CP children who were between the ages of 4 and 6 years
* spasticity grades were 1 and 1+ according to modified Ashworth Scale
* gross motor function classification system at level II and III

Exclusion Criteria:

* Children who have visual impairments, hearing damage
* received Botulinum Toxin injections or oral antispasticity medications within the past 6 months
* fixed deformities at lower limbs
* inability to understand the task

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2025-04-10 (Actual); Primary Completion 2025-07-20 (Actual); Study Completion 2025-09-01 (Actual)

PRIMARY OUTCOMES:
cadence | 8 weeks
  investigators measure cadence
step length and width | 8 weeks
  investigators measure step length, width
gait velocity | 8 weeks
  investigators measure gait velocity
gait time | 8 weeks
  investigators measure gait time
foot angle | 8 weeks
  investigators measure foot angle

CONTACTS AND LOCATIONS:
Overall Officials: mostafa ali, professor, Principal Investigator — associate professor for pediatrics
Locations (1):
- Cairo university, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Undecided